CLINICAL TRIAL: NCT00097851
Title: Phase II Trial of Docetaxel With PI-88 in Patients With Advanced Non-Small-Cell Lung Cancer
Brief Title: Trial of PI-88 With Docetaxel in Advanced Non-Small-Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cellxpert Biotechnology Corp. (Industry)
Collaborators: Medigen Biotechnology Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR88202
Record Dates: First submitted 2004-11-30; First posted 2004-12-01 (Estimated); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: second-line; combination; chemotherapy; anti-angiogenic
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; phosphomannopentaose sulfate

INTERVENTIONS:
Drug: docetaxel
Drug: PI-88

SUMMARY:
PI-88 is a new experimental drug that inhibits tumour growth by reducing the formation of new blood vessels into tumours. Docetaxel is a standard second-line treatment offered to patients with non-small-cell lung cancer who haven't responded to first-line therapies (platinum-based drugs or radiotherapy). Of this group of patients, only 20% remain progression-free 6 months after starting docetaxel treatment. The PR88202 study has been designed to compare two different cancer treatments (docetaxel only, and docetaxel plus PI-88) and to work out which is more effective against the cancer. It is hoped that the combination of PI-88 with docetaxel will allow patients to extend the time it takes for their disease to progress, and also to improve their quality of life.

DETAILED DESCRIPTION:
PR88202 is an open-label randomized study. In the initial phase of the study, patients will be randomized to receive weekly docetaxel alone, or PI-88 in combination with weekly docetaxel. Both groups will receive docetaxel (30 mg/m2), administered by intravenous infusion on days 1, 8 and 15 of a 28-day cycle. The second group only will receive PI-88 (250 mg/day) in addition to docetaxel; PI-88 will be administered by subcutaneous injection on days 1-4, 8-11 and 15-18 of each cycle. The primary efficacy endpoint is the non-progression rate at 6 months. In the extension phase of the study, patients in the combination arm who have stable disease or an objective response after up to six treatment cycles will remain on PI-88 alone as maintenance therapy. Patients who initially receive docetaxel alone and who have disease progression or unacceptable toxicity before the completion of six cycles will be eligible to receive PI-88 alone as third-line therapy.

ELIGIBILITY:
Inclusion Criteria:

* histologically or cytologically confirmed stage IIIb or IV NSCLC that has progressed during or after first-line treatment
* measurable disease by spiral CT chest scan, as defined in RECIST criteria
* performance status 0-1 (ECOG)
* life expectancy at least 2 months
* adequate hemopoietic, renal and hepatic function

Exclusion Criteria:

* current symptomatic central nervous system (CNS) involvement
* prior or co-existent malignancies
* significant non-malignant disease
* acute or chronic gastrointestinal (GI) bleeding in last two years
* inflammatory bowel disease
* abnormal bleeding tendency
* patients at risk of bleeding due to open wounds or planned surgery
* clinically significant hemoptysis within the past 4 weeks
* bilirubin > upper limit of normal (ULN)
* ALT and AST > 2.5 times ULN, or > 1.5 times ULN if alkaline phosphatase > 2.5 times ULN
* alkaline phosphatase > 5 times ULN, unless patient has bone metastases
* myocardial infarction, stroke or congestive heart failure within last 3 months
* prior treatment with docetaxel
* concomitant treatment with aspirin (>100 mg/day), NSAIDs (except selective COX-2 inhibitors, warfarin (>1 mg/day), heparin, LMWH, anti-platelet drugs, CYP3A4 inhibitors
* women who are pregnant or breast-feeding
* women of child-bearing potential not using adequate contraception
* history of allergy and/or hypersensitivity to anti-coagulants or thrombolytic agents, especially heparin
* history of immune-mediated thrombocytopenia, thrombotic thrombocytopenic purpura or other platelet disease
* allergy to polysorbate 80 (component of Taxotere®)
* uncontrolled or serious infection in last 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2004-02; Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Progression-free survival

SECONDARY OUTCOMES:
Time to progression
Response rate
Quality of life
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Nick Pavlakis, MD, Study Chair — Royal North Shore Hospital; Paul Mitchell, MD, Study Director — Austin and Repatriation Hospital
Locations (13):
- Australia (13):
  - Sydney Cancer Centre, Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Sydney Haematology and Oncology Clinics, Hornsby, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Newcastle Mater Misericordiae Hospital, Waratah, New South Wales
  - Prince Charles Hospital, Chermside, Queensland
  - Nambour General Hospital, Nambour, Queensland
  - Mater Hospital, South Brisbane, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - The Queen Elizabeth Hospital, Woodville, South Australia
  - The Alfred Hospital, Prahran, Victoria
  - Border Medical Oncology, Wodonga, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia